CLINICAL TRIAL: NCT00487188
Title: Phase IIIb/IV Randomized, Controlled Study Evaluating an Intensification Treatment Strategy of Adding Enfuvirtide (ENF) to an Oral Highly Active AntiRetroviral Therapy (HAART) in Treatment Experienced Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of Adding Enfuvirtide to Oral Highly Active Antiretroviral Therapy (HAART) in Human Immunodeficiency Virus (HIV) Patients With Prior Treatment Experience
Acronym: INTENSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV18406
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (2):
- ENF + HAART (Experimental): Participants received Enfuvirtide (ENF) 90 mg administered by subcutaneous injection twice a day for up to 48 weeks in addition to an oral highly active antiretroviral treatment (HAART) regimen for up to 48 weeks.
  Interventions: Drug: Enfuvirtide; Drug: Highly active antiretroviral treatment (HAART)
- HAART (Active Comparator): Participants received an oral highly active antiretroviral treatment (HAART) regimen, consisting of 3-5 antivirals for up to 48 weeks.
  Interventions: Drug: Highly active antiretroviral treatment (HAART)

INTERVENTIONS:
Drug: Enfuvirtide — 90 mg subcutaneous injection twice a day
  Other Names: Fuzeon
  Arms: ENF + HAART
Drug: Highly active antiretroviral treatment (HAART) — An oral HAART regimen of 3-5 antiretrovirals was chosen by the physician and patient, based on the patient's prior treatment history and genotypic antiretroviral resistance testing.

SUMMARY:
To assess the efficacy of enfuvirtide (Fuzeon) added to HAART compared to treatment with HAART alone in achieving and maintaining viral load suppression.

DETAILED DESCRIPTION:
This study consisted of two phases. In the Induction phase patients were randomized at Baseline 1 (BL1) in a 1:2 ratio to receive:

* I1: HAART or
* I2: Enfuvirtide (90 mg twice a day) + HAART.

Participants who achieved viral suppression < 50 copies/mL by week 24, confirmed by week 28 or earlier, qualified to enter the Maintenance Phase which started at Baseline 2 (BL2), four weeks after confirmation of response. The Maintenance Phase consisted of three treatment groups:

* M1: HAART continued (patients from I1)

Patients on ENF+HAART (I2) were re-randomized (at a 1:1 ratio) at BL2 to:

* M2: Enfuvirtide stopped and HAART continued
* M3: Enfuvirtide + HAART continued.

The duration of the Maintenance Phase was from BL2 up to 48 weeks after BL1. BL2 could start at the earliest at Week 12 and at the latest Week 32.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults >=18 years of age;
* currently on antiretroviral (ARV) therapy;
* previously treated with 2 or 3 different antiretroviral classes;
* HIV-1 Ribonucleic acid (RNA) >=1,000 copies/mL;
* Cluster differentiation antigen four (CD4) lymphocyte count >=200 cells/mm^3;
* females of childbearing potential must be willing to use a reliable form of effective barrier contraception for the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* history of prior use of enfuvirtide or T-1249;
* women who are pregnant, breastfeeding or planning to become pregnant during the study;
* active, untreated opportunistic infection;
* patients on treatment interruption, or patients interrupting ARV therapy within 4 weeks of screening or during the screening period for reasons either than toxicity management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (3):
  - Cleveland, Ohio
  - Austin, Texas
  - Dallas, Texas
- Vancouver, British Columbia, Canada
- France (5):
  - Le Kremlin-Bicêtre
  - Nantes
  - Paris
  - Poitiers
  - Villeneuve-sur-Lot
- Germany (4):
  - Berlin
  - Bonn
  - Erlangen
  - Frankfurt am Main
- Ramat Gan, Israel
- Italy (5):
  - Bagno a Ripoli
  - Bari
  - Brescia
  - Milan
  - Roma
- Mexico City, Mexico
- Netherlands (2):
  - Amsterdam
  - Tilburg
- Spain (9):
  - Barcelona
  - Cadiz
  - Córdoba
  - Donostia / San Sebastian
  - Huelva
  - Madrid
  - Málaga
  - Seville
  - Valencia
- Zurich, Switzerland

REFERENCES:
- [Derived] Clotet B, Capetti A, Soto-Ramirez LE, Gatell JM, Rowell L, Salgo M, Schapiro JM. A randomized, controlled study evaluating an induction treatment strategy in which enfuvirtide was added to an oral, highly active antiretroviral therapy regimen in treatment-experienced patients: the INTENSE study. J Antimicrob Chemother. 2008 Dec;62(6):1374-8. doi: 10.1093/jac/dkn377. Epub 2008 Sep 8. PMID 18782780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 patients were enrolled into the study at 20 investigational sites in France, Italy, Spain, Mexico, Germany and the US. Study starting 15NOV2005 and ending 5NOV2007.
Pre-assignment Details: In the Induction Phase participants were randomized (2:1 ratio) to receive ENF + HAART or HAART. In the Maintenance Phase participants in the HAART group who responded (viral load < 50 copies/mL) continued to receive HAART; those who responded in the ENF + HAART group were re-randomized (1:1 ratio) to receive ENF + HAART or HAART (ENF removed).
Groups:
- ENF + HAART: Participants received enfuvirtide 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment during the Induction and Maintenance Phase for up to 48 weeks of treatment.
- HAART: Participants received highly active antiretroviral treatment during the Induction and Maintenance Phase for up to 48 weeks of treatment.
- HAART (ENF Removed): Participants who had received ENF + HAART during the Induction Phase and responded to treatment by Week 24 continued to receive HAART alone during the Maintenance Phase, for a total of 48 weeks of treatment.
Period: Induction Phase
Arm/Group | ENF + HAART | HAART | HAART (ENF Removed)
Started | 31 | 16 | 0 (Participants were only randomized to this treatment arm in the Maintenance Phase)
Safety Population | 29 | 18 (2 patients randomized to ENF + HARRT only received treatment with HAART) | 0
Completed | 22 | 9 | 0
Not Completed | 9 | 7 | 0
Not completed — Abnormality of Laboratory Test | 0 | 1 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Refused Treatment | 1 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Administrative | 0 | 1 | 0
Period: Maintenance Phase
Arm/Group | ENF + HAART | HAART | HAART (ENF Removed)
Started | 10 | 8 | 9
Completed | 7 | 8 | 8
Not Completed | 3 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Administrative | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ENF+HAART: Participants received enfuvirtide 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment.
- HAART: Participants received highly active antiretroviral treatment.
- Total: Total of all reporting groups
Arm/Group | ENF+HAART | HAART | Total
Number analyzed (Participants) | 29 | 18 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (7.04) | 41.9 (10.57) | 43.3 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Suppression: HIV-1 RNA < 50 Copies/mL During the Induction Phase
Description: Participants whose viral load achieved suppression (HIV-1 RNA < 50 copies/mL) at Week 24 at the latest, confirmed at Week 28 (2 consecutive assessments ≥ 28 days apart) were defined as responders. Patients who discontinued the study or did not respond to assigned treatment by week 28 were considered as non-responders.
Time Frame: From Baseline 1 to Week 28
Population: Intent-to-Treat Population 1 (ITT1) population (patients evaluable for efficacy in the induction phase)
Measure: Number; unit: Participants
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
Participants | 20 | 8

2. Secondary Outcome: Time to Achieving HIV-1 RNA < 50 Copies/mL During the Induction Phase
Description: The time to achieving HIV-1 RNA <50 copies/mL was counted from Baseline 1 until the first of the two consecutive <50 copies/mL measurements.
  Patients who discontinued from the study or patients who did not have confirmed virological response by week 28 were classed as non-responders and censored at Week 24.
Time Frame: Baseline 1 until Week 28.
Population: Intent-to-Treat Population 1 (ITT1) population (patients evaluable for efficacy in the induction phase).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
days | 57.0 [29 to 119] | 141.0 [70 to NA] — The 75% quartile could not be calculated as >75% of patients did not achieve HIV-1 RNA < 50 Copies/mL in this arm.

3. Secondary Outcome: Number of Participants With Viral Suppression HIV-1 RNA < 400 Copies/mL During the Induction Phase
Description: Participants whose viral load achieved suppression (HIV-1 RNA < 400 copies/mL) by Week 24 at the latest, confirmed at Week 28 (2 consecutive assessments ≥ 28 days apart) were defined as responders. Patients who discontinued the study or did not respond to assigned treatment by Week 28 were considered as non-responders.
Time Frame: From Baseline 1 to Week 28
Population: ITT1 population (patients evaluable for efficacy in the induction phase)
Measure: Number; unit: Participants
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
Participants | 21 | 8

4. Secondary Outcome: Change From Baseline to Week 24 in Viral Load
Description: Change from Baseline in log10 HIV-1 RNA at Week 24. Least squares means were calculated from an analysis of covariance (ANCOVA) model with treatment, a flag variable "removed ENF at re-randomization" and Baseline viral load as independent variables.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat Population 1 (ITT1) population (patients evaluable for efficacy in the Induction Phase). Baseline values were carried forward (i.e. the change from baseline set to zero) for patients with missing data at week 24 or who withdrew prior to the week 24 time window.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
log10 copies/mL | -1.402 (0.69) [-1.854 to -0.949] | -1.156 (0.61) [-1.710 to -0.601]

5. Secondary Outcome: Change From Baseline to Week 24 in Cluster Differentiation Antigen Four Positive (CD4+) Cell Counts
Description: Change from Baseline in CD4+ Cell Counts at Week 24. Least squares means were calculated from an ANCOVA model with treatment as an independent variable.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
cells/mm^3 | 20.81 [-18.89 to 60.50] | 17.88 [-37.38 to 73.13]

6. Secondary Outcome: Percentage of Induction Phase Participants With Viral Load < 50 Copies/mL at 48 Weeks
Description: The percentage of participants from the Induction Phase who maintained HIV-1 RNA < 50 Copies/mL at Week 48. Patients who discontinued from the study, rebounded to ≥ 50 copies/mL (i.e., had two consecutive readings ≥ 50 copies/mL), had missing data or had virological failure by Week 48 were classed as non-responders.
Time Frame: Week 48
Population: Induction Phase Intent-to-Treat Population 1 (ITT1).
Measure: Number; unit: percentage of participants
Groups:
- ENF+HAART: Participants received enfuvirtide (ENF) 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment (HAART) in the Induction Phase. In the Maintenance Phase, participants either continued to receive ENF+HAART or HAART alone.
  This group contains all patients who were randomized to ENF+HAART at BL1 and follows the patients throughout 48 weeks, regardless of which arm they were randomized to at BL2.
- HAART: Participants received highly active antiretroviral treatment during both the Induction and Maintenance Phase.
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 31 | 16
percentage of participants | 45.2 | 25.0

7. Secondary Outcome: Percentage of Maintenance Phase Participants With Viral Load < 50 Copies/mL at 48 Weeks
Description: The percentage of participants from the Maintenance Phase who maintained HIV-1 RNA < 50 copies/mL at Week 48. Patients who discontinued from the study, rebounded to ≥ 50 copies/mL (i.e., had two consecutive readings ≥ 50 copies/mL), had missing data or had virological failure by Week 48 were classed as non-responders.
Time Frame: Week 48
Population: Maintenance Phase Intent-to-Treat Population 2 (ITT2).
Measure: Number; unit: percentage of participants
Groups:
- ENF+HAART: Participants received enfuvirtide (ENF) 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment (HAART) in the Induction Phase. In the Maintenance Phase, participants either continued to receive ENF+HAART or HAART alone.
  This group contains all patients who entered the Maintenance phase from the ENF+HAART Induction phase, regardless of which arm they were randomized to at BL2.
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 19 | 8
percentage of participants | 73.7 | 50.0

8. Secondary Outcome: Change From Baseline to Week 48 in Cluster Differentiation Antigen Four Positive (CD4) Cell Counts
Description: Change from Baseline in CD4 Cell Counts at Week 48. Least squares means were calculated from an ANCOVA model with treatment and baseline CD4 count as independent variables.
Time Frame: Baseline 1 and Week 48
Population: Intent-to-Treat Population 2 (ITT2) population (patients evaluable for efficacy in the Maintenance Phase). Baseline values were carried forward (i.e. the change from baseline set to zero) for patients with missing data at week 48 or who withdrew prior to the week 48 time window.
Measure: Least Squares Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 19 | 8
cells/mm^3 | 73.09 [-4.10 to 150.28] | 50.79 [-68.24 to 169.83]

9. Secondary Outcome: Time to Loss of Viral Response During the Maintenance Phase
Description: The time to loss of viral response (defined as HIV-1 RNA <50 copies/mL) was counted from Baseline 2 until the first of two consecutive ≥50 copies/mL measurements.
  Only patients who were qualified for entering the Maintenance Phase were included in the analysis.
Time Frame: From Baseline 2 to Week 48.
Population: Maintenance Phase Intent-to-Treat Population 2 (ITT2)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 19 | 8
days | NA [NA to NA] — Median time to loss of viral response could not be estimated due to the low number of patients with loss of viral response in this arm (4 out of 19 ITT2 patients) and the inter-quartile range was not calculated. | NA [NA to NA] — Median time to loss of viral response could not be estimated due to the low number of patients with loss of viral response in this arm (3 out of 8 ITT2 patients) and the inter-quartile range was not calculated.

10. Secondary Outcome: Time to Virological Failure During the Maintenance Phase
Description: Time to virological failure (defined as HIV-1 RNA ≥ 400 copies/mL) was counted from Baseline 2 until the first of the two consecutive ≥400 copies/mL measurements.
  Only patients who were qualified for entering the Maintenance Phase were included in the analyses.
Time Frame: From Baseline 2 to Week 48.
Population: Maintenance Phase Intent-to-Treat Population 2 (ITT2)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 19 | 8
days | NA [NA to NA] — Median time to virological failure could not be estimated due to the low number of patients with virological failure in this arm and the inter-quartile range was not calculated. | NA [NA to NA] — Median time to virological failure could not be estimated due to the low number of patients with virological failure in this arm and the inter-quartile range was not calculated.

11. Secondary Outcome: Number of Participants With Virological Failure During the Maintenance Phase
Description: Virological failure was defined by 2 consecutive HIV-1 RNA values ≥ 400 copies/mL during the Maintenance Phase.
Time Frame: From Baseline 2 to Week 48.
Population: Maintenance Phase Intent-to-Treat Population 2 (ITT2)
Measure: Number; unit: Participants
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 19 | 8
Participants | 3 | 0

12. Secondary Outcome: Percentage of Participants Maintaining CD4+ Count During the Maintenance Phase
Description: Maintenance of CD4+ count defined as having greater than or equal to 200 cells/mm^3 at Baseline 2 (BL2) and greater than or equal to 200 cells/mm^3 at Week 48.
Time Frame: Baseline 2 to Week 48.
Population: Maintenance Phase ITT2 population with a Baseline 2 CD4+ count of greater than or equal to 200 cells/mm^3.
Measure: Number; unit: percentage of participants
Arm/Group | ENF + HAART | HAART | HAART (ENF Removed)
Number analyzed (Participants) | 9 | 8 | 8
percentage of participants
  Week 48 CD4+ Count ≥200 cells/mm^3 | 66.67 | 75.00 | 75.00
  Week 48 CD4+ Count Missing | 33.33 | 25.00 | 12.50

13. Secondary Outcome: Percentage of Participants With Improvement in CD4+ Count During the Maintenance Phase
Description: Improvement of CD4+ count defined as having from 100 to less than 200 CD4+ cells/mm^3 at Baseline 2 (BL2) and greater than or equal to 200 cells/mm^3 at Week 48.
Time Frame: Baseline 2 to Week 48.
Population: Maintenance Phase ITT2 population with a Baseline 2 CD4+ count of ≥100 to <200 cells/mm^3.
Measure: Number; unit: percentage of participants
Arm/Group | ENF + HAART | HAART | HAART (ENF Removed)
Number analyzed (Participants) | 1 | 0 | 1
percentage of participants
  Week 48 CD4+ Count ≥200 cells/mm^3 | 100.00 |  | 100.00
  Week 48 CD4+ Count Missing | 0 |  | 0

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) During the Induction Phase
Description: A serious AE (SAE) is an event which: results in death, is life-threatening, disabling or incapacitating; is a congenital anomaly in the offspring of a patient who received study drug; requires or prolongs inpatient hospitalization; jeopardizes the patient or require medical or surgical intervention to prevent one of the outcomes above; any Grade 4 laboratory value considered by the investigator clinically significant or that requires an action; any injection site reaction that meets SAE criteria above. Non-serious AEs reported include pneumonia and non-serious AEs that led to discontinuation.
Time Frame: Start of the study treatment until the end of the Induction Phase (Week 12 to Week 32)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ENF+HAART | HAART
Number analyzed (Participants) | 29 | 18
participants
  Serious Adverse Event | 3 | 3
  Non-serious Adverse Event | 3 | 1
  Adverse Events Leading to Withdrawal | 5 | 1

ADVERSE EVENTS:
Time Frame: From the start of the study treatment until 28 days after the last dose of the study medication.
Description: Per protocol, AEs of pneumonia (non-serious and serious), AEs that lead to discontinuation, and AEs that are serious were reported. Unless fatal, any acquired immunodeficiency syndrome (AIDS)-defining events (ADEs), as defined by the 1993 Center for Disease Control (CDC) AIDS Surveillance Case Definitions, are excluded from the definition of SAE.
Groups:
- Induction: ENF+HAART: During the Induction Phase participants received enfuvirtide 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment for a maximum of 32 weeks.
- Induction Phase: HAART: During the Induction Phase participants received highly active antiretroviral treatment for a maximum of 32 weeks.
- Maintenance Phase: ENF + HAART: During the Maintenance Phase, participants who had received ENF+HAART and who responded to treatment during the Induction Phase continued to receive enfuvirtide 90 mg subcutaneously twice a day in combination with highly active antiretroviral treatment for up to 48 weeks of total treatment.
- Maintenance Phase: HAART (ENF Removed): During the Maintenance Phase, participants who had received ENF+HAART and who responded to treatment during the Induction Phase continued to receive HAART alone during the Maintenance Phase, for up to a total of 48 weeks treatment.
- Maintenance Phase: HAART: During the Maintenance Phase, participants who had received HAART alone and who responded to treatment during the Induction Phase continued to receive highly active antiretroviral treatment for up to 48 weeks of total treatment.
Arm/Group | Induction: ENF+HAART | Induction Phase: HAART | Maintenance Phase: ENF + HAART | Maintenance Phase: HAART (ENF Removed) | Maintenance Phase: HAART
Serious Adverse Events (participants affected / at risk) | 3/29 | 3/18 | 2/10 | 3/9 | 0/8
Other Adverse Events (participants affected / at risk) | 9/29 | 11/18 | 2/10 | 4/9 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: ENF+HAART (N=29) | Induction Phase: HAART (N=18) | Maintenance Phase: ENF + HAART (N=10) | Maintenance Phase: HAART (ENF Removed) (N=9) | Maintenance Phase: HAART (N=8)
PAROTITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: ENF+HAART (N=29) | Induction Phase: HAART (N=18) | Maintenance Phase: ENF + HAART (N=10) | Maintenance Phase: HAART (ENF Removed) (N=9) | Maintenance Phase: HAART (N=8)
DIARRHOEA (Gastrointestinal disorders) | 2 | 5 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1 | 1 | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
GINGIVAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 2 | 0 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
ABSCESS JAW (Infections and infestations) | 0 | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ONYCHOMYCOSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 1 | 0 | 0 | 0
SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.